CLINICAL TRIAL: NCT06305104
Title: Phase 2 Clinical Trial of Randomized, Blinded, Positive-controlled to Explore the Skin Test Dosage of EEC in People Aged 18 to 65 Years Old and the Safety and Preliminary Efficacy in People Aged 3 to 75 Years Old.
Brief Title: Clinical Trial to Explore the Skin Test Dosage of EEC in People Aged 18 to 65 Years Old and the Safety and Preliminary Efficacy in People Aged 3 to 75 Years Old.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu CoenBiotech Co., Ltd (Industry)
Collaborators: Beijing Chest Hospital, Capital Medical University (Other); Wuhan Institute for Tuberculosis Control (Other); The Public Health Clinical Center of Chengdu (Unknown); Xuzhou Infectious Disease Hospital (Unknown); Jiangsu Province Centers for Disease Control and Prevention (Network); Changde First People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KN-EEC-II
Record Dates: First submitted 2024-01-16; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- TB subjects in 18-65 years old (Experimental): 140 TB subjects's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC,2.5 μg /ml or 5 μg /ml ) and the control drug (inoculated in both arms of the same body); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 2.5μg/ml EEC; Biological: 5μg/ml EEC; Biological: 5 unit（U） EC
- healthy subjects in 18-65 years old (Experimental): 180 healthy subjects's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC,2.5 μg /ml or 5 μg /ml ) and the control drug (inoculated in both arms of the same body); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 2.5μg/ml EEC; Biological: 5μg/ml EEC; Biological: 5 unit（U） EC
- non-TB subjects with lung disease in 18-65 years old (Experimental): 40 non-TB subjects with lung disease in 18-65 years old,each subject's left and right arms were randomly assigned to receive a single intradermal injection of 0.1 ml of the test drug (EEC,2.5 μg /ml or 5 μg /ml ) and the control drug (inoculated in both arms of the same body); all subjects were intradermally injected into the middle and lower 1/3 of the volar side of the forearm using the Mantoux method. injection. The time between skin tests on the left and right arms must be at least 30 minutes (skin test on the left arm first, then on the right arm). The follow-up visit observation point is based on the completion time of the second dose of injection.
  Interventions: Biological: 2.5μg/ml EEC; Biological: 5μg/ml EEC; Biological: 5 unit（U） EC
- TB subjects in 3-17 years old and 66-75 years old (Experimental): Each enrolled subject received a single intradermal injection of 0.1 ml of the test drug (EEC) in one arm; the Mantoux method was used to inject intradermally into the middle and lower 1/3 of the volar side of the forearm.
  Interventions: Biological: 5μg/ml EEC
- non-TB subjects in 3-17 years old and 66-75 years old (Experimental): Each enrolled subject received a single intradermal injection of 0.1 ml of the test drug (EEC) in one arm; the Mantoux method was used to inject intradermally into the middle and lower 1/3 of the volar side of the forearm.
  Interventions: Biological: 5μg/ml EEC

INTERVENTIONS:
Biological: 2.5μg/ml EEC — 0.1ml ,one time, containing low dose of 2.5μg/ml of active ingredients
  Arms: TB subjects in 18-65 years old; healthy subjects in 18-65 years old; non-TB subjects with lung disease in 18-65 years old
Biological: 5μg/ml EEC — 0.1ml, one time, containing high dose 5μg/ml of active ingredients
Biological: 5 unit（U） EC — 0.1 ml , one time, containing 5U of active ingredients
  Arms: TB subjects in 18-65 years old; healthy subjects in 18-65 years old; non-TB subjects with lung disease in 18-65 years old

SUMMARY:
This is a randomized, blind, positive-controlled study to explore the skin test dosage of recombinant mycobacterium tuberculosis fusion protein ( EEC) in the population aged 18 to 65 years old , and to further evaluate the safety and preliminary efficacy of EEC in the population aged 3 to 75 years old.

In the first stage,180 healthy subjects, 140 tuberculosis（TB）subjects and 40 non-TB subjects with lung diseases aged 18 to 65 years old are divided into different groups through a randomized, blind methods. Every group carry out a low-dose (2.5μg/ml) or high-dose (5μg/ml) study, with 180 subjects in each dose group .Every subject injects intradermally EEC and EC randomly in both arms of the same person. Evaluate the consistency of assay results of EEC, EC and Interferon-Gamma Release Assay（IGRA）.Evaluate the sensitivity, specificity and consistency of assay results of EEC, EC and IGRA in healthy people, TB patients and non-TB patients with lung diseases, and determine the optimal dose of EEC for clinical auxiliary diagnosis of tuberculosis.

In the second stage, 60 healthy subjects and TB subjects aged 3-17 years and 66-75 years old are divided into different groups through a randomized, open, single-arm method with the target dose. Evaluate the safety, tolerance and preliminary efficacy of target dose of EEC in healthy people and TB patients aged 3 to 17 years old and 66 to 75 years old.

DETAILED DESCRIPTION:
In the first stage,180 healthy subjects, 140 TB subjects and 40 non-TB subjects with lung diseases which meet the standard respectively are divided into different groups through a randomized blind methods.Every group carry out a low-dose (2.5μg/ml) or high-dose (5μg/ml) study, with 180 subjects in each dose group.

Each subject's left and right arms will be randomly assigned to receive an intradermal injection of the experimental drug EEC and the control drug inoculated in both arms of the same person. A drug(EEC or EC) is injected in left arm first, observe 30 min and if no obvious adverse reaction ,then another drug (EEC or EC) will be injected in right arm. Observe and record the vital signs (breathing, heart rate, blood pressure ,temperature),the skin specific reaction (diameters of flush and induration of injection site) at 24h, 48h, 72h, 96h, and 7 days after skin test;local reactions (redness, pain, swelling, rash,itching) and a variety of adverse events. Evaluate the sensitivity , specificity and consistency rate of assay results of EEC, EC and IGRA in healthy subjects, TB patients and non-TB patients with lung diseases,determine the optimal dose of EEC for clinical auxiliary diagnosis of tuberculosis,and further evaluate the safety of EEC in healthy subjects, TB patients and non-TB patients with lung diseases.

In the second stage, 60 subjects aged 3-17 years old (30 cases) and 66-75 years old (30 cases) are enrolled, including 30 healthy subjects and 30 TB patients. Every subject is divided into different groups through a randomized, open label method, and receive a single intradermal injection of experimental drug (EEC) in one arm. Observe and record the vital signs (breathing, heart rate and temperature); laboratory examination and electrocardiogram (ECG) ;the skin specific reactions of injection site at 4h,8h,24h, 48h, 72h, 96h, and 7 days after skin test ; local reactions and a variety of adverse events，to further evaluate the safety and preliminary efficacy of EEC in people aged 3 to 75 years old.

ELIGIBILITY:
Inclusion Criteria:

* For healthy subjects:

  1. At the time of enrollment - For healthy subjects:enrollment is 3 ~ 75 years old (including 3 years old and 75 years old), regardless of gender ;
  2. Guardians of persons aged 3-7 years , persons aged 8-17 years old and their guardians, persons aged 18-75 years old themselves and/or their guardians (spouse or children) agree to participate in this trial and sign an informed consent form;
  3. The person and/or guardian can comply with the requirements of the clinical trial protocol to participate in /accompany the subject to follow- up visits;
  4. After medical history inquiry, there is no history of tuberculosis (including intrapulmonary and external tuberculosis ) and close contact history with tuberculosis patients (referring to direct contact with registered tuberculosis patients from 3 months before diagnosis to 14 days after starting anti-tuberculosis treatment);
  5. Those who have no clinical symptoms of tuberculosis poisoning and whose chest imaging examination (for subjects aged 15 to 75 years old) is normal or abnormal without clinical significance;
  6. Normal or abnormal measurements of vital signs ( axillary temperature, pulse , respiration , blood pressure ) and electrocardiogram have no clinical significance; [ The axillary temperature of all subjects was measured < 37.3°C ; blood pressure was measured in subjects aged 18-75 years (systolic blood pressure <160 millimetres of mercury（mmHg） and diastolic blood pressure <100mmHg) ; pulse and respiration were determined by the researcher based on the subject's age]
  7. Physical examinations are normal or abnormal with no clinical significance;
  8. Laboratory tests including blood routine, urine routine, and blood biochemistry tests were all normal or abnormal with no clinical significance.
* For patients with tuberculosis (including pulmonary tuberculosis):

  1. Those who was diagnosed with tuberculosis/ pulmonary tuberculosis according to the "People's Republic of China Health Industry Standard Pulmonary Tuberculosis Diagnostic Criteria " combined with the "Technical Guidelines for Tuberculosis Prevention and Control in China ( 2021 Edition )" (accepted clinical comprehensive analysis diagnosis);
  2. The age at the time of enrollment is 3 to 75 years old (including 3 years old and 75 years old), regardless of gender ;
  3. Guardians of persons aged 3-7 years old, persons aged 8-17 years old and their guardians, persons aged 18-75 years old themselves and/ or their guardians (spouse or children) agree to participate in this trial and sign an informed consent form;
  4. The person and /or guardian may comply with the requirements of the clinical trial protocol and participate in follow-up visits.
* For patients with non-tuberculous lung disease

  1. Patients with clear clinical diagnosis of pulmonary disease, and the clinician can rule out pulmonary tuberculosis and extrapulmonary tuberculosis based on the patient's clinical manifestations, imaging and laboratory tests (including IGRA );
  2. Age at the time of enrollment is 18 to 65 years old (including 18 years old and 65 years old), regardless of gender;
  3. Those who agree to participate in this trial and sign the informed consent form;
  4. Those who may comply with the requirements of the clinical trial protocol and participate in follow-up visits

Exclusion Criteria:

* Those with known or suspected (or high-risk) severe immune diseases, immune function impairment or abnormalities ( except HIV infection /AIDS ), including:
* who have convulsions, epilepsy, a history of mental illness and / or a family history of mental illness (immediate relatives);
* People with allergies, such as those who have a history of allergies to two or more drugs or foods, or those who are known to be allergic to the components of this medicine;
* Those currently suffering from acute infectious diseases (such as measles, whooping cough, influenza, etc.), acute conjunctivitis, acute otitis media, and generalized skin diseases;
* After consultation, have a history of past or current serious heart, liver, kidney, digestive system, respiratory system, nervous system, mental disorder and metabolic disorders;
* Those who are currently suffering from acute febrile illness; or those who have used antipyretic, analgesic and anti-allergic drugs within 3 days before the skin test and which may affect the research evaluation as assessed by the researcher ;
* People with serious infections (such as pyoderma, severe eczema, etc.);
* who are participating in or participating in any other new drug clinical trials within 3 months;
* Have received non-live vaccines within 7 days before the skin test , or have received live attenuated vaccines within 28 days ;
* Lactating or pregnant women, or female subjects of childbearing age who have a positive pregnancy test before enrollment and who have not taken effective contraceptive measures 2 weeks before enrollment.
* Those with a history of drug abuse;
* Any other circumstances that the investigator believes may affect the evaluation of the study.

Ages: 3 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-07-18 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of different doses of EEC and control EC in pulmonary tuberculosis patients aged 18 to 65 years ; | 7days after injection
  Sensitivity (also known as the true positive rate which is defined as the percentage of actual disease that is correctly judged to be diseased according to the diagnostic criteria of the test)of different doses of EEC and control EC in patients with pulmonary tuberculosis aged 18 to 65 years old.
specificity of different doses of EEC and control EC in healthy subjects aged 18 to 65 years and patients with non-tuberculous lung disease ; | 7days after injection
  Specificity (also known as true negative rate which is defined as the percentage of actual disease-free patients correctly judged to be disease-free according to the diagnostic criteria of the test) of different doses of EEC and control EC in healthy people and patients with non-tuberculous lung disease aged 18 to 65 years old.
The skin test site specific reaction at 4h,8h (only for stage 2);24h, 48h, 72h, 96h, and 7 days after skin test. Those with average diameter of induration/redness is ≥5 mm will be considered to positive. | 7days after injection
  Endpoint of skin test site specific response evaluation which is defined as the skin test site symptom at 4 hour(only for stage 2), 8 hour(only for stage 2）, 24 hour ,48 hour,72 hour,96 hour and 7 days after the skin test such as redness, induration, double ring, blister, necrosis, and lymphangitis (any symptoms of double ring, blister, necrosis, and lymphangitis were strongly positive).

SECONDARY OUTCOMES:
Receiver operator characteristic curve(ROC) of different doses of EEC to evaluate the optimal diagnostic test cut-off value of the test drug. | 7days after injection
Area under the curve(AUC) of different doses of EEC to evaluate the optimal diagnostic test cut-off value of the test drug. | 7days after injection
In healthy people, patients with tuberculosis and patients with non-tuberculous lung diseases, the consistency rates of the three detection reagents EEC , EC and IGRA were evaluated respectively. | 7days after injection
  The consistency rate of EC, EEC and IGRA detection reagents which is defined as the pairwise KAPPA values of the three detection methods in different dose groups among healthy people, patients with pulmonary tuberculosis and patients with non-tuberculosis pulmonary disease( the Kappa values of the three detection methods in different dose groups were calculated respectively ).
Incidence of adverse events and serious adverse events at injection and non-injection sites，abnormal incidence of laboratory indicators and vital signs during the study period. | 7days after injection
  Safety endpoint including: incidence of adverse events at injection and non-injection sites within 7 days after skin test; abnormal incidence of laboratory indicators (blood routine, blood biochemistry, urine routine, ECG test) at 72 hour after skin test; abnormal incidence of vital signs within 7 days after skin test; incidence of serious adverse events after skin test during the study period.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Beijing Chest Hospital, Beijing, Beijing Municipality
  - Wuhan Institute for Tuberculosis Control, Wuhan, Hubei
  - Changde First People's Hospital, Changde, Hunan
  - Jiangsu Province Centers for Disease Control and Prevention, Nanjing, Jiangsu
  - Xuzhou Infectious Disease Hospital, Xuzhou, Jiangsu
  - Public health clinical center of chengdu, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided